CLINICAL TRIAL: NCT02337686
Title: Pharmacodynamic Study of Pembrolizumab in Patients With Recurrent Glioblastoma
Brief Title: Pembrolizumab in Treating Patients With Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0820; NCI-2015-00174 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0820 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-01-08; First posted 2015-01-14 (Estimated); Results first posted 2023-01-11 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Glioblastoma; Recurrent Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, surgery) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day -21 and day -1, and then undergo surgery on day 0. After 2-3 weeks or recovery from surgery, patients continue to receive pembrolizumab IV over 30 minutes every 3 weeks. Courses repeat every 42 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Other: Pharmacological Study; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Pharmacological Study — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase II trial studies the effects of pembrolizumab on the body, or pharmacodynamics, in patients with glioblastoma that has come back. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate immune effector function in resected glioblastoma tissue after treatment with intravenously administered pembrolizumab monotherapy in the neoadjuvant setting in patients with recurrent glioblastoma.

II. To correlate the progression free survival at 6 months (PFS6) with objective increases in the immune effector T cell: regulatory T cell (Treg) ratio in tumor tissue as measured by ex vivo T-cell-specific cytokines profiling.

SECONDARY OBJECTIVES:

I. Comparison of time to progression of last prior therapy to time to progression on pembrolizumab, median duration of response, overall response rate (ORR), and overall survival (OS) and safety.

TERTIARY OBJECTIVES:

I. To identify imaging characteristics associated with immunological changes in tumor following treatment with pembrolizumab.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day -21 and day -1, and then undergo surgery on day 0. After 2-3 weeks or recovery from surgery, patients continue to receive pembrolizumab IV over 30 minutes every 3 weeks. Courses repeat every 42 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Have histologically confirmed World Health Organization grade IV malignant glioma (glioblastoma or gliosarcoma); participants will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of glioblastoma or variants is made
* Patients must be at first or second relapse and clinically require reoperation for tumor progression within 4 to 6 weeks; Note: relapse is defined as progression following initial therapy (i.e., radiation, chemotherapy, or radiation + chemotherapy); if the participant had a surgical resection for relapsed disease and no anti-tumor therapy instituted for up to 12 weeks, this is considered one relapse; for participants who had prior therapy for a low grade glioma, the surgical diagnosis of a high grade glioma will be considered first relapse
* Have measurable disease consisting of a minimal volume of 1 cm^3
* Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion
* Have a performance status of >= 60 on the Karnofsky performance scale (KPS)
* Stable dose of steroids for 5 days, no more than 2 mg dexamethasone (or equivalent) total per day
* Absolute neutrophil count (ANC) >= 1,500/mcL (performed within 14 days prior to registration)
* Platelets >=100,000/mcL (performed within 14 days prior to registration)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (performed within 14 days prior to registration)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (performed within 14 days prior to registration)
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (performed within 14 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases (performed within 14 days prior to registration)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (performed within 14 days prior to registration)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (performed within 14 days prior to registration)
* Female subject of childbearing potential should have a negative serum pregnancy test
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Has been treated previously with bevacizumab
* Has tumor localized primarily to the brainstem or spinal cord
* Has received prior interstitial brachytherapy, implanted chemotherapy, or therapeutics delivered by local injection or convection enhanced delivery
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device 4 weeks since last dose of agent administration
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy > 2 mg of dexamethasone total per day or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent; Note: subjects with alopecia, =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known carcinomatous meningitis, extracranial disease, or multifocal disease
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-programmed cell death (PD)-1, anti-PD ligand (PD-L)1, anti-PD-L2, anti-cluster of differentiation (CD)137 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies); testing not required
* Has known history of hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected); testing not required
* Has received a live vaccine within 30 days prior to the first dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Puduvalli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] de Groot J, Penas-Prado M, Alfaro-Munoz K, Hunter K, Pei BL, O'Brien B, Weathers SP, Loghin M, Kamiya Matsouka C, Yung WKA, Mandel J, Wu J, Yuan Y, Zhou S, Fuller GN, Huse J, Rao G, Weinberg JS, Prabhu SS, McCutcheon IE, Lang FF, Ferguson SD, Sawaya R, Colen R, Yadav SS, Blando J, Vence L, Allison J, Sharma P, Heimberger AB. Window-of-opportunity clinical trial of pembrolizumab in patients with recurrent glioblastoma reveals predominance of immune-suppressive macrophages. Neuro Oncol. 2020 Apr 15;22(4):539-549. doi: 10.1093/neuonc/noz185. PMID 31755915
- See also: MD Anderson Cancer Center — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants recruited at MD Anderson Cancer Center.
Pre-assignment Details: A total of 18 participants were consented; 3 screen failures.
Groups:
- Treatment (Pembrolizumab, Surgery): 200 mg, intravenously (IV) once every 3-weeks prior to surgery for two doses and then restarting 200 mg Q 2-wk following surgical resection
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Surgery)
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Surgery)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival at 6 Months
Description: Progression-free survival, defined as the time from study enrollment until the time of first occurrence of disease progression, relapse, or death due to disease. Patients who are alive without progression or relapse will be censored at the time of last contact. Response Assessment in Neuro-Oncology (RANO) Criteria for Evaluating Response.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Surgery)
Number analyzed (Participants) | 15
Participants | 15

2. Secondary Outcome: Number of Participants With Progression
Description: Defined as the length of time from the date of diagnosis or the start of treatment for a disease until the disease starts to get worse or spread to other parts of the body. Time to Progression measured by the method of Kaplan and Meier.
Time Frame: The time from study enrollment until the time of first occurrence of disease progression, relapse, or death due to disease, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Surgery)
Number analyzed (Participants) | 15
Participants | 10

3. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Surgery)
Number analyzed (Participants) | 15
months | 20 [8.64 to 28.45]

4. Secondary Outcome: Number of Participants With Response Rate
Description: Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate. Per the Response Assessment in Neuro-Oncology (RANO) Criteria for Evaluating Response for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=50% decrease in the sum of the products of perpendicular diameter of measurable lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Surgery)
Number analyzed (Participants) | 14
Participants | 3

5. Secondary Outcome: Number of Adverse Events
Description: Adverse events as defined by the Common Terminology Criteria for Adverse Events (CTCAE) version 4 for grades 1, 2, and 3. There were no grade 4 AEs.
Time Frame: Up to 30 days after completion of study treatment
Measure: Number; unit: number of adverse events
Arm/Group | Treatment (Pembrolizumab, Surgery)
Number analyzed (Participants) | 15
number of adverse events
  Adverse Event Grade 1 | 31
  Adverse Event Grade 2 | 18
  Adverse Event Grade 3 | 6

ADVERSE EVENTS:
Time Frame: adverse events will be recorded from the baseline through 30 days following the end of treatment and at each examination. Serious adverse events will be collected for 90 days after the end of treatment. All-Cause Mortality will be assessed for up to 2 years.
Arm/Group | Treatment (Pembrolizumab, Surgery)
All-Cause Mortality (participants affected / at risk) | 14/15
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pembrolizumab, Surgery) (N=15)
Hydrocephalus (Nervous system disorders) | 5
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 3
Edema cerebral (Nervous system disorders) | 1
Wound dehiscence (Nervous system disorders) | 1
Neoplasms benign malignant and unspecified (incl and polyps (other) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Enterocolitis infections (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pembrolizumab, Surgery) (N=15)
Fatigue (General disorders) | 12
Gait disturbance (Musculoskeletal and connective tissue disorders) | 4
Dysphasia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Urinary tract Infection (Renal and urinary disorders) | 1
Edema face (Infections and infestations) | 2
Pain Extremity (Musculoskeletal and connective tissue disorders) | 1
Lung Infection (Infections and infestations) | 1
Otitis Media (Ear and labyrinth disorders) | 1
Tremor (Musculoskeletal and connective tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Chill (General disorders) | 1
Insomia (Psychiatric disorders) | 2
Anorexia (Gastrointestinal disorders) | 2
Pruritius (Skin and subcutaneous tissue disorders) | 2
General muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
Ataxia (Musculoskeletal and connective tissue disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Fever (General disorders) | 1
Flushing (Vascular disorders) | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 1
Hyperthyroidism (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Memory Impairment (Nervous system disorders) | 2
Urinary Frequency (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Fatigue (General disorders) | 2
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT02337686/Prot_SAP_000.pdf